CLINICAL TRIAL: NCT06505629
Title: Paired Emotion Reading Improves Emotion Regulation in Rural Children With Adverse Childhood Experiences: A Cluster Randomized Controlled Trial
Brief Title: Paired Emotion Reading Improves Emotion Regulation in Rural Children With ACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Paired Reading in ACE Children
Record Dates: First submitted 2024-07-04; First posted 2024-07-17 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Emotion Regulation; Adverse Childhood Experience
Keywords: Emotion Regulation; Randomized Controlled Trial; Adverse Childhood Experience; Children; Mental Health
MeSH Terms: conditions — Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the online Paired Emotion Reading Intervention (PERI) (Experimental)
  Interventions: Behavioral: the online Paired Emotion Reading Intervention (PERI)
- the online Paired General Reading Intervention (PGRI) (Active Comparator)
  Interventions: Behavioral: the online Paired General Reading Intervention (PGRI)
- Care as Usual (CAU) (No Intervention)

INTERVENTIONS:
Behavioral: the online Paired Emotion Reading Intervention (PERI) — In the PERI, all children will receive three books about emotion knowledge. The paired reading groups will read and discuss these books over the next six weeks. Before starting the reading sessions, the paired groups will meet online via video to get to know each other and set reading goals. During the reading process, participants will check in daily with their reading progress. From the second week to the fifth week, participants will engage in weekly online discussions about the reading content. These discussions, led by the urban children, will follow a semi-structured discussion guide. The discussions aim to deepen the children's understanding of the book content and facilitate the application of emotion-related knowledge and emotion regulation strategies in their daily lives. The discussion sessions will be recorded and uploaded for regular review by the researchers.
  Arms: the online Paired Emotion Reading Intervention (PERI)
Behavioral: the online Paired General Reading Intervention (PGRI) — Apart from the differences in the reading materials and discussion topics, all other aspects are identical to the PERI group. In the online PGRI, children will read three books of their choice, and discussions will center around general reading experiences and feelings.
  Arms: the online Paired General Reading Intervention (PGRI)

SUMMARY:
The goal of this study is to explore the feasibility and effectiveness of the online Paired Emotion Reading Intervention (PERI) on the emotion regulation of rural children with adverse childhood experiences (ACE), as compared with the online Paired General Reading Intervention (PGRI) group and a Care as Usual (CAU) control group. This study is a cluster randomized controlled trial and will recruit three rural schools, randomly assigning them to PERI, PGRI, or CAU. Each school will recruit 50 children with ACE. Additionally, the investigators will recruit 150 urban children of similar ages to the rural children. Urban and rural children will be randomly paired to form urban-rural reading groups, reading different types of books and engaging in discussions. It is hypothesized that, after the intervention, rural children in the PERI group will show significantly greater improvements in emotion regulation self-efficacy and emotional awareness compared to the PGRI and CAU groups. These group differences are expected to persist at 1-month and 3-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria for rural children:

1. Age between 9 and 15 years;
2. Experience of at least one adverse childhood experience;
3. Independent reading ability in Chinese;
4. Could use electronic devices such as mobile phones, tablets, or computers for online paired reading;
5. Informed consent obtained from both the child and their parents.

Exclusion Criteria for rural children: A past or current diagnosis of a mental disorder.

The inclusion and exclusion criteria for urban children are the same, except they do not need to meet criterion 2.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Emotional awareness of rural children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  The investigators explored the effectiveness of PERI on the emotional awareness of rural children using the Emotional Awareness Questionnaire (EAQ). The EAQ consists of 30 items, each rated on a 3-point scale, with higher scores indicating greater emotional awareness.
Emotion regulation self-efficacy of rural children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  The investigators explored the effectiveness of PERI on the emotion regulation self-efficacy of rural children using the modified subscale of the Emotional Self-Efficacy Scale. Each item is rated on a 5-point scale, with higher scores indicating higher self-efficacy in emotion regulation.

SECONDARY OUTCOMES:
Mental health symptoms of rural children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  The investigators examined the effectiveness of PERI on the mental health of rural children using the Strengths and Difficulties Questionnaire (SDQ), including both parent-report and child-report versions, along with three items from the Children's Depression Inventory (CDI) measuring feelings of loneliness. The SDQ comprises five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Relationship Problems, and Prosocial Behavior. Each subscale consists of 5 items rated on a scale of 0-2. Higher scores on each subscale indicate greater difficulties, except for the Prosocial Behavior subscale. Higher score on the items of CDI indicates higher level of loneliness.
Resilience of rural children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  The investigators explored the effectiveness of PERI on the resilience of rural children through the 10-item Connor-Davidson Resilience Scale. Each item is rated on a 5-point scale, with higher scores indicating higher level of resilience.
Self-esteem of rural children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  The investigators explored the effectiveness of PERI on the self-esteem of rural children through the Rosenberg self-esteem scale. The total score ranges from 0 to 30, with higher scores indicating greater self-esteem.
Emotional awareness of urban children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  Urban children will complete the Emotional Awareness Questionnaire (EAQ), as rural children did. The EAQ consists of 30 items, each rated on a 3-point scale, with higher scores indicating greater emotional awareness.
Emotion regulation self-efficacy of urban children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  Urban children will complete the modified subscale of the Emotional Self-Efficacy Scale, as rural children did. Each item is rated on a 5-point scale, with higher scores indicating higher self-efficacy in emotion regulation.
Mental health symptoms of urban children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  The investigators examined the effectiveness of PERI on the mental health of urban children using the Strengths and Difficulties Questionnaire (SDQ), including both parent-report and child-report versions, along with three items from the Children's Depression Inventory (CDI) measuring feelings of loneliness. The SDQ comprises five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Relationship Problems, and Prosocial Behavior. Each subscale consists of 5 items rated on a scale of 0-2. Higher scores on each subscale indicate greater difficulties, except for the Prosocial Behavior subscale. Higher score on the items of CDI indicates higher level of loneliness.
Resilience of urban children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  Urban children will complete the 10-item Connor-Davidson Resilience Scale. Each item is rated on a 5-point scale, with higher scores indicating higher level of resilience.
Self-esteem of urban children | baseline, post treatment (6 weeks), 10 weeks, 18 weeks
  Urban children will complete the Rosenberg self-esteem scale.The total score ranges from 0 to 30, with higher scores indicating greater self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided